CLINICAL TRIAL: NCT05598034
Title: Optimization of tDCS Brain Network Engagement in Depression
Brief Title: Evaluating tDCS Brain-stimulation in Depression Using MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mayank Anant Jog, Postdoctoral Scholar, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MH128572; K99MH128572 (NIH)
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Major Depressive Disorder
Keywords: Transcranial Direct Current Stimulation (tDCS); MRI; Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Left DLPFC tDCS (Experimental): Participants randomized to this arm will receive tDCS at the left DLPFC brain region.
  Interventions: Device: Left DLPFC tDCS
- Left DLPFC tDCS + task (Experimental): Participants randomized to this arm will receive tDCS at the left DLPFC brain region. Additionally, participants will be asked to perform a mental task (2-back working memory) at the same time.
  Interventions: Device: Left DLPFC tDCS; Behavioral: Cognitive task
- Right DLPFC tDCS (Experimental): Participants randomized to this arm will receive tDCS at the right DLPFC brain region.
  Interventions: Device: Right DLPFC tDCS
- Right DLPFC tDCS + task (Experimental): Participants randomized to this arm will receive tDCS at the right DLPFC brain region. Additionally, participants will be asked to perform a mental task (2-back working memory) at the same time.
  Interventions: Device: Right DLPFC tDCS; Behavioral: Cognitive task

INTERVENTIONS:
Device: Left DLPFC tDCS — This intervention involves placing non-invasive scalp-electrodes over the left DLPFC brain region to deliver a mild, tolerable electric current.
  Arms: Left DLPFC tDCS; Left DLPFC tDCS + task
Device: Right DLPFC tDCS — This intervention involves placing non-invasive scalp-electrodes over the right DLPFC brain region to deliver a mild, tolerable electric current.
  Arms: Right DLPFC tDCS; Right DLPFC tDCS + task
Behavioral: Cognitive task — Participants will be asked to perform a 2-back working memory mental task alongside administered tDCS
  Arms: Left DLPFC tDCS + task; Right DLPFC tDCS + task

SUMMARY:
Patients, physicians, and those who fund depression research are keenly interested in depression treatments that do not involve taking medications. One promising candidate treatment is transcranial direct current stimulation (tDCS), a low-cost technique that involves placing electrodes on specific scalp locations and using a 9-volt battery to cause a small amount of electricity to pass through parts of the brain. Depending on the direction of electrical flow, tDCS can make brain cells (neurons) more likely or less likely to generate their own electrical signals. When evaluated as a treatment, tDCS is typically done in daily sessions over a period of two weeks.

One of the challenges of tDCS is to work out the best possible positioning of electrodes and direction of electricity flow to gradually cause lasting changes in brain activity in ways that might be expected to improve depression. To address this challenge, the investigators are using MRI to take pictures of the brain during tDCS. This data will help us better understand the short-term effects of tDCS in depression and help us learn how to customize future treatments to cause a lasting beneficial response.

Patients with depression between the ages of 20-55 years are eligible to take part in this research. Potential participants will undergo:

1. An assessment to confirm eligibility. This will take place over a secure videoconference call lasting no more than 3 hours.
2. Two in-person study visits lasting 30 min and 2-1/2 hours respectively. In the first visit, the investigators will use the MRI to take a picture of the brain and head structure to determine appropriate locations for placing the tDCS electrodes at the start of the second visit. Following electrode placement, an MRI scan will be performed to take pictures of the brain during tDCS. Depending on the study arm,

   1. Participants may receive 'active' or 'sham' tDCS. The 'sham' condition is identical to the 'active' tDCS in every way except that it involves minimal tDCS and is designed to help rule out effects unrelated to the administered tDCS electricity.
   2. Participants may also be asked to perform a mental task during MRI.

All participants will be compensated $150 + parking upon completion of all study-visits.

DETAILED DESCRIPTION:
Depression is characterized by disruption in the regulation of emotion and mood. Converging evidence from multiple brain imaging studies indicates that depression is associated with dysfunction in the top-down, emotion-regulating frontoparietal brain regions that include the hypoactive left dorsolateral prefrontal cortex (DLPFC) brain region and the hyperactive right DLPFC. Dysfunction in additional brain regions including the cingulate cortex, hippocampus and amygdala has also been linked to depressive symptoms. Together, these brain regions form the dorso-fronto-limbic brain network, and beneficial modulation of this specific network has been hypothesized to improve depressive symptoms.

Network modulation is feasible using a wide range of brain stimulation techniques, including transcranial direct current stimulation (tDCS). The latter technique has recently received high interest in the context of moderate depression due to its demonstrated safety, low-cost and non-invasive nature. A typical tDCS setup consists of non-invasive electrodes placed on the scalp to administer tolerable electric currents at specific brain targets. The administered electric current has been shown to modulate brain activity depending on the direction of the applied electricity, with anodal tDCS increasing neuronal activity at the brain-target, and cathodal tDCS decreasing activity at the targeted brain region. Consequently, tDCS setups in depression have typically targeted the aforementioned hypoactive left DLPFC using anodal tDCS and/or the hyperactive right DLPFC using cathodal tDCS. However, the downstream effects of tDCS on the dorso-fronto-limbic network are not fully understood. Understanding the engagement of this depression-relevant brain network by tDCS could provide important insights into optimizing tDCS setups for antidepressant applications. Consequently, the current study is proposing to use MRI techniques to map and investigate network engagement by tDCS in depression, as described below. Note that while Study arm 1 will use data from an existing study, arms 2-4 will involve recruitment of depressed participants de-novo.

1. Study arm 1 will investigate the engagement of the dorso-fronto-limbic brain network in depression when 'active' or 'sham' anodal tDCS is administered at the left DLPFC brain region at rest. 'Sham' tDCS provides a control condition to facilitate the measurement of tDCS-specific effects, and besides involving minimal electricity, is designed to be identical to 'active' tDCS in every other way (e.g. electrode placement, etc.). For this arm, de-identified data from an ongoing clinical trial in depression with separate aims will be acquired for analysis (NCT04507243, N=48 participants, randomized to 24 'active' and 24 'sham' groups).
2. Study arm 2 will investigate network engagement when anodal tDCS is administered at the left DLPFC brain region during the performance of a mental task (2-back working memory). N=24 subjects will be enrolled using a single group experimental design incorporating a within-session control condition (instead of a separate 'sham' group as in Arm 1). Participation will involve one assessment over a secure videoconference call to confirm eligibility (lasting no more than 3 hours), and two in-person study visits (lasting 30 min and 2.5 hours respectively). Both in-person visits will involve MRI's: the first visit's MRI scans will help determine tDCS electrode positioning for the second visit, and the second visit's MRI scans will help us map changes in brain activity and connectivity during tDCS.
3. Study arms 3 and 4 will investigate network engagement during right DLPFC cathodal tDCS. N=48 participants will be recruited for arm 3 (randomized to 24 'active' and 24 'sham') and N=24 participants will be recruited for arm 4. In all other respects, study arms 3 and 4 will be identical to study arms 1 and 2 respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 20 to 55 years, inclusive
2. Gender: all
3. Race/ethnicity: all races and ethnic groups
4. Capacity to provide informed consent
5. Hamilton Rating Scale for Depression score of ≥17 and <24, with or without symptoms of anxiety.
6. Treatment naïve or on a stable standard antidepressant regimen (including selective serotonin reuptake inhibitors (SSRIs), serotonin-noradrenaline reuptake inhibitors (SNRIs), monoamine oxidase inhibitors (MOAIs) or tricyclic's (TCAs)) with no change in treatment 6-weeks prior to and during the tDCS intervention.
7. Work at UCLA or live within 1-hr driving distance of UCLA

Exclusion Criteria:

1. Pregnancy
2. Non-English speaking (due to scales administered)
3. Substance Use Disorder within last 12 months
4. Neurological condition associated with brain abnormalities (e.g., traumatic brain injury; recent stroke, tumor)
5. Any contraindication to tDCS (e.g., skin disease or treatment causing irritation)
6. Any condition that would contraindicate scanning (metal implants, claustrophobia or a breathing or movement disorder)
7. Currently receiving any form of psychotherapy
8. Change in antidepressant medication within 6-weeks of starting the trial
9. Severe or treatment resistant depression - HAMD scores > 24 and a history of a major depressive episode lasting >2- years or failure to 2 or more antidepressant trials in the current index episode
10. Any neuromodulation therapy (e.g., ECT, rTMS, DBS, VNS or tDCS) within the last 3-months
11. Current or past (within the last 1-month) use of anticonvulsants, lithium, psychostimulant, dexamphetamine
12. Current use of decongestants or other medication previously shown to interfere with cortical excitability
13. Diagnosis: Schizophrenia Axis I disorder, or dementia of any type
14. Bipolar I disorder (due to possible risk of mania and because lithium and anticonvulsants are excluded).
15. On regular benzodiazepine medication that it is not clinically appropriate to discontinue for the 2-week duration of the trial
16. Depression related to serious medical illness (i.e., mood disorder due to general medical condition) 17. Actively suicidal as defined by a score of 4 on item 3 of HAMD

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Activity changes in the dorso-fronto-limbic brain network | Within the 2.5 hour fMRI session
  fMRI-BOLD signal within nodes of the dorso-fronto-limbic brain network will be analyzed for activity changes concurrent with tDCS

SECONDARY OUTCOMES:
Connectivity changes in the dorso-fronto-limbic brain network | Within the 2.5 hour fMRI session
  fMRI-BOLD signal within nodes of the dorso-fronto-limbic brain network will be analyzed for connectivity changes occuring with tDCS

CONTACTS AND LOCATIONS:
Overall Officials: Mayank A Jog, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No